CLINICAL TRIAL: NCT04505033
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HB0017 Following a Single Dose in Adult Healthy Volunteers
Brief Title: A Study of Injection HB0017 in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HB0017-01
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- 50 mg s.c (Experimental)
  Interventions: Drug: HB0017
- 50 mg placebo (Placebo Comparator)
  Interventions: Drug: placebo
- 150 mg s.c. (Experimental)
  Interventions: Drug: HB0017
- 150 mg placebo (Placebo Comparator)
  Interventions: Drug: placebo
- 300 mg s.c. (Experimental)
  Interventions: Drug: HB0017
- 300 mg placebo (Placebo Comparator)
  Interventions: Drug: placebo
- 450 mg s.c. (Experimental)
  Interventions: Drug: HB0017
- 450 mg placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HB0017 — HB0017 at 100 mg/mL (1 mL/vial) in 2 mL glass vial with a rubber stopper. HB0017 will be administered in the abdominal area by a subcutaneous injection in the mornings. A maximum volume of 1 mL is injected per site.
  Other Names: recombinant humanized IgG1 monoclonal antibody
  Arms: 150 mg s.c.; 300 mg s.c.; 450 mg s.c.; 50 mg s.c
Drug: placebo — A matching injection solution containing a specific volume of normal saline (0.9%, Sodium Chloride Injection USP) and no active substance will be prepared for the subjects who will be assigned to placebo according to the dose schedule.
  Other Names: 0.9%, Sodium Chloride Injection USP
  Arms: 150 mg placebo; 300 mg placebo; 450 mg placebo; 50 mg placebo

SUMMARY:
placebo by subcutaneous (SC) administration. Forty subjects (10 subjects per cohort for SC administration) will be randomized and assigned to up to 4 sequential doses cohorts of HB0017 (50 mg, 150 mg, 300 mg and 450 mg) or matching placebo. Each cohort of ten volunteers will be randomly assigned to receive either a single dose of HB0017 or matching placebo at a ratio of 4:1. Starting with the lowest dose, each of the subsequent doses will be administered only if the preceding dose was determined to be safe and well tolerated. The decision to escalate the next dose will be made jointly by the sponsor s medical expert and the investigator based upon review of 15-day blinded safety data prior to dosing each cohort.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects must meet the following criteria to be eligible for study entry:

1. Healthy male or female subjects age ≥ 18 and ≤ 55 years.
2. Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized since at least 6 months) must be willing to use one of the following acceptable contraceptive method throughout the study and for 112 days after the study drug administration:

   * Simultaneous use of intra-uterine contraceptive device without hormone release system placed at least 4 weeks prior to study drug administration, and condom for the male partner;
   * Simultaneous use of diaphragm with intravaginally applied spermicide and male condom for the male partner, starting at least 21 days prior to study drug administration.
3. Male subjects who are not vasectomized for at least 6 months, and who are sexually active with non-sterile female partner [sterile female partners include post-menopausal women (absence of menses for 12 months prior to drug administration) or women who have had a tubal ligation, hysterectomy, or bilateral oophorectomy (at least 6 months prior to drug administration)] must be willing to use one of the following acceptable contraceptive method throughout the study and for 112 days after the study drug administration:

   * simultaneous use of condom, and for the female partner hormonal contraceptives (used since at least 4 weeks) or intra-uterine contraceptive device (placed since at least 4 weeks);
   * simultaneous use of male condom, and for the female partner, diaphragm with intravaginally applied spermicide;
4. Body Mass Index (BMI) ≥ 18.5 and ≤ 30 kg/m².
5. No clinically significant findings in the medical history and physical examination.
6. No clinically significant laboratory values (including urinalysis), unless the investigator considers any abnormality to not be clinically significant.
7. Normal ECG, blood pressure, respiratory rate, temperature and heart rate, unless the investigator considers any abnormality to be not clinically significant.
8. Informed consent must be obtained in writing for all subjects enrolled into the study.

Exclusion Criteria:

-

Subjects who meet any of the following criteria will be excluded from study entry:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease.
2. Current or history of malignancy (subjects with squamous cell skin cancer maybe included based on investigator assessment.).
3. Family history of premature Coronary Heart Disease (CHD).
4. Treatment in the previous 3 months with any drug known to have a well-defined potential for toxicity to a major organ. Exposure to any prescription medication 14 days prior to randomization, to herbal remedies or over-the counter medications 7 days prior to randomization.
5. Participation in another research with any investigational product within 28 days or 5 half-lives of the drug, whichever is greater, before screening.
6. Any medical history of asthma, allergic rhinitis or urticarial, or any other clinically significant allergy reaction including food allergy. Known allergy to biologics.
7. Blood or plasma donation of more than 500 mL during the previous 2 months and/or more than 50 mL in the 2 weeks prior to screening.
8. Had a vaccination with a live attenuated vaccine within 6 months prior to dosing.
9. Subjects at risk for tuberculosis (TB), specifically subjects with:

   * Current clinical, radiographic or laboratorial evidence of active TB.
   * History of active tuberculosis or exposure to endemic areas within 8 weeks prior to QuantiFERON®-TB testing performed at screening.
   * Positive QuantiFERON®-TB test with positive chest X-ray, indicating possible tuberculosis infection. Subjects with positive QuantiFERON®-TB test with documented completion of treatment for latent TB can be included into the study.
10. Positive test for hepatitis B, hepatitis C, or HIV at screening.
11. History of clinically significant opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia).
12. Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to screening.
13. Presence of fever (body temperature > 37.6°C) (e.g., a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to the first dosing.
14. History of drug abuse within 1 year prior to screening, or use of soft drugs (such as marijuana) within 3 months prior to the screening, or hard drugs (such as cocaine, phencyclidine, and crack) within 1 year prior to screening. Positive drug screen(cocaine, methamphetamine, phencyclidine, and Tetrahydrocannabinol) at screening or Day -1.
15. History of regular alcohol consumption exceeding 14 drinks/week for female subjects or 21 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening. Positive Breath Alcohol Test at screening or Day -1.
16. Current cigarette smoker (cigarettes or e-cigarettes) who smoke over 5 cigarettes per day within 3 months prior to screening.
17. Mental condition rendering the subject incapable of understanding the nature, scope, and possible consequences of the study.
18. Pregnant or Breasting feeding subject. Positive pregnancy test (HCG) within 3 days prior to Day 1.
19. Adults under guardianship and people with restriction of freedom by administrative and legal decisions.
20. Unlikely to comply with the clinical study protocol; e.g. uncooperative attitude, inability to return for followed-up visit, and improbability of completing the study.
21. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 113Days.
  Incidence, nature, relatedness, and severity of AEs.

SECONDARY OUTCOMES:
AUC (Area Under Curve) after single dose | 1month
  AUC (Area Under Curve) after single dose
T1/2 (Elimination Half-life) after single dose | 1month
  T1/2 (Elimination Half-life) after single dose
Cmax (Maximum Serum Concentration) after single dose | 1 month
  Cmax (Maximum Serum Concentration) after single dose

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland Clinical Studies Ltd, Grafton, Auckland, New Zealand

REFERENCES:
- [Derived] Jiang C, Du Y, Liu X, Wang J, Ge C, Xu J, Wang S, Li B, Zhu G, Zhang W, Qian Q, Ma C, Zhu X, Zhan Y, Yang Y. Safety, tolerability, pharmacokinetics and efficacy of HB0017, a humanized monoclonal antibody that targets interleukin-17A, in healthy participants and patients with moderate-to-severe plaque psoriasis. Br J Dermatol. 2023 Dec 20;190(1):28-36. doi: 10.1093/bjd/ljad315. PMID 37669307